CLINICAL TRIAL: NCT00821600
Title: Single-Dose, Open-Label Pilot Study to Explore the Pharmacokinetics, Safety and Tolerability of a Gluteal Intramuscular Injection of a 4-Week Long-Acting Injectable Formulation of Risperidone in Patients With Chronic Stable Schizophrenia
Brief Title: Characterization of Intramuscular Injections of Risperidone 4 Week Long-acting Injectable (LAI) Formulation in the Buttock of Patients With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015742
Record Dates: First submitted 2009-01-09; First posted 2009-01-13 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Psychotic Disorders; Schizophrenia
Keywords: Risperidone; Antipsychotic; Pharmacokinetic; Long-acting Injectable
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 001 (Experimental): risperidone IR and LAI formulation 1 mg risperidone IR single injection followed after 7 to 14 days with 75mg risperidone 4-week-LAI single injection
  Interventions: Drug: risperidone IR and LAI formulation

INTERVENTIONS:
Drug: risperidone IR and LAI formulation — 1 mg risperidone IR single injection, followed after 7 to 14 days with 75mg risperidone 4-week-LAI single injection

SUMMARY:
The purpose of this study is to explore the pharmacokinetics, safety and tolerability of a 4-week long-acting injectable (LAI) formulation of risperidone after single intramuscular (i.m.) injection of 75 mg risperidone LAI in the gluteal muscle.

DETAILED DESCRIPTION:
An intramuscular injectable formulation of risperidone long-acting formulation is under development with the aim to provide a sustained and stable level of risperidone during each treatment cycle given every 4 weeks. As this formulation is a long acting formulation, patients will be treated with a 1 mg immediate release (IR) formulation in the first week to confirm that the patient does not develop an allergic reaction to the drug before receiving the long acting injectable (LAI) formulation. Each patient receives a total of two injections. The first one is the immediate release formulation and the second one, which is given at least a week later, is the new long acting formulation. Eligible patients can stay on their previous oral medication, no tapering of medication is needed. Blood samples will be collected to determine the levels of risperidone and its major metabolite in plasma. Blood samples will be obtained by venipuncture (needle stick) immediately before (pre-dose) and at 5, 10, 20, 30, 45 min, 1, 1.5, 2, 4, 6, 8,12, 16, 24, 36, 48, 72, 96 hours after the 1st injection and at 2, 6, 12, 24, 48, 96 hrs, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 34, 36, 39, 43, 50, 57, 64, 71, 78, 85 days after the second injection of risperidone. Safety will assessed at visits throughout the study by monitoring scores of the Clinical Global Impression - Severity (CGI-S), scores of Extrapyramidal Symptom Rating Scale (ESRS), adverse events (AE), changes in clinical laboratory results, changes in physical examinations (PE), changes in electrocardiograms (ECGs), as well as patient and investigator evaluation of the injection site. The study has two periods. In the first period all patients will receive one injection of 1 mg risperidone IR (immediate release) solution (liquid). The follow-up duration is 96 hours. In the second period, patients will receive one injection of risperidone 4-week formulation of 75 mg. The follow-up duration is 85 days. The injections, administered in the muscle of the buttocks, will be given 7 to 14 days apart.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of schizophrenia
* Clinically stable with no change in current antipsychotic medications
* Meet Positive and Negative Symptom Score (PANSS) and Clinical Global Impression (CGI) score criteria
* Have a body mass index (BMI) between 18 and 35 kilogram (kg)/meter (m)2
* If a woman, is postmenopausal surgically sterile, abstinent, or, if sexually active, is practicing before entry into the study and agrees to practice throughout the study an effective method of birth control
* If a man, agrees to use an adequate contraception method as deemed appropriate by the investigator

Exclusion Criteria:

* Alcohol or substance dependence, with the exception of nicotine or caffeine dependence
* Involuntarily-committed or unable to provide an informed consent
* Has tardive dyskinesia, History of Neuroleptic Malignant Syndrome
* History of or current clinically significant medical illness
* Treatment with any protocol disallowed therapies
* Clinically significant result from screening laboratory or ECG

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To explore the pharmacokinetics of a 4-week long acting injectable (LAI) formulation of risperidone after single intramuscular (IM) injection of 75 mg in the gluteal muscle. | Up to 85 days for 4-week LAI formulation of risperidone and up to 96 hrs for immediate release (IR) formulation

SECONDARY OUTCOMES:
To explore safety and tolerability of a 4-week LAI formulation of risperidone by monitoring scores on CGI-S, scores on ESRS, AEs, PE, lab values, ECG values and injection site reactions. | Up to 85 days

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (3):
- United States (3):
  - Cerritos, California
  - Santa Ana, California
  - Atlanta, Georgia

REFERENCES:
- See also: Single Dose, Open Label Pilot Study to Explore the Pharmacokinetics, Safety and Tolerability of a Gluteal Intramuscular Injection of a 4 Week Long Acting Injectable Formulation of Risperidone in Subjects With Chronic Stable Schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=797&filename=CR015742_CSR.pdf